CLINICAL TRIAL: NCT04537871
Title: Cardiovascular Reserve Evaluation in Survivors of Transplantation (CREST)
Brief Title: Cardiovascular Reserve Evaluation in Survivors of Transplant, CREST Study
Status: Active, not recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19424; NCI-2020-06749 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19424 (Other: City of Hope Medical Center); P30CA033572 (NIH); R01HL150069 (NIH)
Record Dates: First submitted 2020-08-27; First posted 2020-09-03 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Hematopoietic and Lymphoid Cell Neoplasm; Hodgkin Lymphoma; Myelodysplastic Syndrome; Non-Hodgkin Lymphoma; Plasma Cell Myeloma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Hematologic Neoplasms; Hodgkin Disease; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin; Multiple Myeloma | interventions — Exercise Test; Clostridium perfringens epsilon-toxin; Respiratory Physiological Phenomena; High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (physical assessment): Patients undergo echocardiogram to assess cardiac function and mechanics, cardiopulmonary exercise test, pulmonary function test, musculoskeletal ultrasound, bioelectrical impedance analysis to measure total lean body mass and percent body fat), physical function tests, and collection of blood samples within 45 days from the start of conditioning therapy, and at 6 months, 1 year, and 2 years post-transplant.
  Interventions: Procedure: Bioelectric Impedance Analysis; Procedure: Biospecimen Collection; Procedure: Cardiopulmonary Exercise Testing; Procedure: Echocardiography; Procedure: Physical Performance Testing; Procedure: Pulmonary Function Test; Other: Questionnaire Administration; Procedure: Ultrasound

INTERVENTIONS:
Procedure: Bioelectric Impedance Analysis — Undergo bioelectric impedance analysis
  Other Names: BIA; Bioelectric Impedance; Bioelectric Impedance Test; Bioelectrical Impedance Analysis; Bioimpedance Analysis
Procedure: Biospecimen Collection — Undergo collection of blood samples
Procedure: Cardiopulmonary Exercise Testing — Undergo cardiopulmonary exercise test
  Other Names: CPET; CPX
Procedure: Echocardiography — Undergo echocardiogram
Procedure: Physical Performance Testing — Undergo physical function tests
  Other Names: Physical Fitness Testing; Physical Function Testing
Procedure: Pulmonary Function Test — Undergo pulmonary function test
  Other Names: lung function test; PFT; Pulmonary Function Testing; Pulmonary Function Tests
Other: Questionnaire Administration — Ancillary studies
Procedure: Ultrasound — Undergo musculoskeletal ultrasound

SUMMARY:
This study evaluates how well the heart, lungs, and muscles are working individually, and how these systems are working together in transplant survivors. Information collected in this study may help doctors to understand why hematopoietic stem cell transplant survivors are at higher risk for developing cardiovascular disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate cardiovascular reserve capacity, as measured by peak oxygen consumption (VO2peak), in hematopoietic cell transplantation (HCT) survivors.

II. Define the determinants of VO2peak impairment in HCT survivors.

OUTLINE:

Patients undergo echocardiogram to assess cardiac function and mechanics, cardiopulmonary exercise test, pulmonary function test, musculoskeletal ultrasound, bioelectrical impedance analysis to measure total lean body mass and percent body fat), physical function tests, and collection of blood samples within 45 days from the start of conditioning therapy, and at 6 months, 1 year, and 2 years post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* Age at HCT >= 18 years
* Diagnosis of acute leukemia (myeloid, lymphoid), lymphoma (non-Hodgkin, Hodgkin), multiple myeloma or myelodysplastic syndromes
* Planning to undergo first autologous or allogeneic transplant
* Able to fluently read and write in English
* Able to understand and sign the study specific informed consent form (ICF)
* Physically able and willing to complete all study procedures

Exclusion Criteria:

* Unstable bone lesions per electronic medical record review and/or notification from patient's primary physician
* Unstable angina or history of acute myocardial Infarction (< 5 days of any planned study procedures)
* Recurrent syncope
* Acute myocarditis or pericarditis
* Symptomatic severe aortic stenosis
* Uncontrolled arrhythmia causing symptoms
* Pulmonary embolus < 3 month of study procedures
* Thrombosis of lower extremities
* Moderate or severe persistent asthma (National Asthma Education & Prevention)
* Room air desaturation at rest =< 85%
* Non-cardiopulmonary disorders that may affect exercise performance or be aggravated by exercise (i.e. infection, renal failure, thyrotoxicosis)
* Anemia (hemoglobin [Hgb] < 8 g/dL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute leukemia (myeloid, lymphoid), lymphoma (non-Hodgkin, Hodgkin), multiple myeloma or myelodysplastic syndromes
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular reserve capacity, as measured by VO2peak, in HCT survivors | Up to 24 months post-hematopoietic cell transplantation (HCT)
  We will measure initial VO2peak in patients prior to HCT and its post-HCT trajectory over time; compare VO2peak in HCT survivors at baseline (pre-HCT), 6m, 1Y, and 2Y post-HCT to established age- and sex-normative data; and define the association between VO2peak and self-reported health-related quality of life (HRQOL) at baseline/over time.
Determinants of VO2peak impairment in HCT survivors | Up to 24 months post-hematopoietic cell transplantation (HCT)
  We will use Generalized Estimating Equation(GEE) and generalized linear models to examine the correlation between VO2peak and measures of:
  1. cardiac (left ventricular function/ contractility [systolic, diastolic, cardiac output, strain], ventricular-arterial (VA) coupling, arterial elastance);
  2. pulmonary (obstructive, restrictive lung disease, diffusion capacity);
  3. musculoskeletal (body composition [% lean muscle mass], muscle quality, two minute step in place test, 30 second sit to stand test, timed up and go); and
  4. hematologic function, adjusting for potential confounding variables (e.g. age, sex) and time since HCT.

CONTACTS AND LOCATIONS:
Overall Officials: Saro H Armenian, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-11): https://cdn.clinicaltrials.gov/large-docs/71/NCT04537871/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-08): https://cdn.clinicaltrials.gov/large-docs/71/NCT04537871/ICF_001.pdf